CLINICAL TRIAL: NCT05365997
Title: Behavioral Nudges to Improve Palliative Care Utilization in Advanced Cancer
Acronym: BE-EPiC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UPCC 29921; 849498 (Other: UPenn IRB)
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Cancer
Keywords: Cancer; Palliative Care; Behavioral Economics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Each clinician pod will be randomized in a 1:1 fashion to either intervention or usual care.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Clinicians will receive no further interventions beyond usual practice.
- Intervention (Experimental): Clinicians receive a nudge consisting of an electronic health record in-basket message indicating a patient has a default pended order for palliative care.
  Interventions: Other: Default Nudge

INTERVENTIONS:
Other: Default Nudge — For patients whose clinician pods are randomized to the intervention arm, the care team pod will receive a message indicating that the patient is eligible for palliative care and that a default referral order has been pended for that patient. Clinicians will be given an opportunity to respond if they do not want their patient to be referred to palliative care. For clinicians who do not respond, after the allotted time, the Clinical Research Coordinator will reach out to the patient to introduce palliative care and ask if staff can schedule an appointment. For clinicians who respond no, the pended order will be removed and no patient contact by the research team will occur.
  Arms: Intervention

SUMMARY:
Patients with cancer often undergo costly therapy and acute care utilization that is discordant with their wishes, particularly at the end of life. Despite early palliative care consultations being a National Comprehensive Cancer Network (NCCN) guideline-concordant practice in advanced cancer, palliative care referral rates for stage IV patients are low. In this project, the investigators will evaluate a health system initiative that uses behavioral nudges to prompt palliative care referrals among outpatients with advanced cancer in terms of successful palliative care referrals and downstream quality of life outcomes. In partnership with the health system, this will be conducted as a 2-arm pragmatic cluster randomized trial.

DETAILED DESCRIPTION:
Patients with advanced cancer have poor quality of life and life expectancy. Palliative care is a medical specialty focusing on providing relief from the symptoms and stress of serious illnesses such as cancer. While palliative care referrals often occur in the inpatient setting for acutely ill individuals, early outpatient specialty palliative care concurrent with cancer-directed treatment improves quality of life and survival, is an evidence-based practice, and is endorsed by national guidelines. Palliative care can be provided in the ambulatory, telemedicine, or home-based settings. However, nearly half of patients with advanced cancer do not receive palliative care prior to dying. Lack of standardized referral criteria and screening methods for palliative care contributes to underutilization. There is a high need for strategies to increase use of palliative care in oncology.

Clinicians underutilize palliative care, initiating referrals a median of 2 months before death. This status quo bias, which predisposes clinicians to continue current practice even if not the optimal option, may lead to delayed or missed palliative care referrals. Additionally, optimism bias, the cognitive bias that causes clinicians to believe that their own patients are at lesser risk of negative outcomes, may cause clinicians to underestimate a patient's mortality risk or symptom burden, thus delaying palliative care referral. Finally, overconfidence bias, the propensity to overestimate one's desired behaviors when it is not objectively reasonable, may lead clinicians to incorrectly believe they are initiating more palliative care referrals than their peers.

Overcoming suboptimal clinician decision-making biases are key to increasing palliative care referrals. Principles from behavioral economics can inform "nudges" that change how clinicians receive information and make choices such as palliative care referral. Default, opt-out nudges that make the optimal choice the path of least resistance can mitigate clinicians' status quo bias. Reframing clinicians' prognoses by providing data-driven life expectancy assessments may combat optimism bias.

Early palliative care intervention can improve quality of life for patients with advanced cancer. Outpatient palliative care is available at 98% of National Cancer Institute (NCI)-designated cancer centers and 63% of non-NCI centers. Early outpatient palliative care concurrent with cancer-directed treatment improves quality of life, reduces symptom burden, and decreases rates of aggressive end of life care. Nevertheless, only a minority of patients who qualify for palliative care receive it.

The primary objective of the study is to evaluate the impact of sending behavioral nudges to clinicians, as compared to usual practice, on completion of palliative care referrals among patients with advanced cancer. Our secondary objectives are to identify the impact of prompted palliative care referrals on quality of life, acute care utilization, and end-of-life utilization. This is a 2-arm pragmatic randomized trial among approximately 250 outpatients with advanced cancer to assess response to behavioral nudges to refer to palliative care. The setting will be outpatient oncology at the Ann B. Barshinger Cancer Institute at Lancaster General Health. Eligible clinicians will be randomized in clusters by overlapping clinical team (pod) to receive default electronic medical record-based prompts for palliative care referral among advanced cancer patients (Arm 1) vs no intervention/usual practice (Arm 2). These nudges have been shown to positively influence clinician behavior and are often used to drive value-based oncology care; however, they have never been studied in the context of palliative care referral. The primary outcome is completion of a palliative care referral within 12 weeks of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Have a functional telephone number
* Receive ongoing care from hematology/oncology services within the Ann B. Barshinger Cancer Institute (ABBCI) at Lancaster General Health.

Exclusion Criteria:

* Patients appearing for a new patient visit
* Patients who have previously received palliative care
* Patients who are enrolled in an ongoing clinical trial of a therapeutic agent
* Patients who receive primary oncologic care within another institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Parikh, MD, MPP, Principal Investigator — Penn/ACC
Locations (1):
- Ann B. Barshinger Cancer Institute at Lancaster General Health, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parikh RB, Sedhom R, Ferrell WJ, Villarin K, Berwanger K, Scarborough B, Oyer R, Kumar P, Ganta N, Sivendran S, Chen J, Volpp KG, Bekelman JE. Behavioural economic interventions to embed palliative care in community oncology (BE-EPIC): study protocol for the BE-EPIC randomised controlled trial. BMJ Open. 2023 Mar 24;13(3):e069468. doi: 10.1136/bmjopen-2022-069468. PMID 36963789

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinician Pod
Groups:
- Control: Usual Care
- Intervention: Nudge group
Period: Overall Study
Arm/Group | Control | Intervention
Started | 136; 2 Clinician Pod | 130; 2 Clinician Pod
Completed | 136; 2 Clinician Pod | 130; 2 Clinician Pod
Not Completed | 0; 0 Clinician Pod | 0; 0 Clinician Pod

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 136 | 130 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (13) | 66 (12.7) | 66.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 147
  Male | 62 | 57 | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 129 | 123 | 252
  Race: Black or African American | 3 | 4 | 7
  Race: Asian | 3 | 0 | 3
  Race: Mixed | 0 | 1 | 1
  Race: Unknown/not reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 3 | 3 | 6
  Ethnicity: non-Hispanic | 133 | 127 | 260
Diagnosis [Count of Participants; unit: Participants]
  CNS | 0 | 1 | 1
  Brain | 1 | 0 | 1
  Head and neck | 3 | 12 | 15
  Thoracic | 0 | 1 | 1
  Lung | 33 | 12 | 45
  Liver | 1 | 0 | 1
  Pancreatic | 4 | 2 | 6
  GI | 17 | 7 | 24
  Colon/rectal/anal | 30 | 16 | 46
  GYN | 1 | 25 | 26
  GU | 4 | 12 | 16
  Breast | 25 | 25 | 50
  Melanoma | 5 | 2 | 7
  Other | 12 | 15 | 27
Advanced Solid Malignancy [Count of Participants; unit: Participants] | 131 | 128 | 259
Brain Metastasis [Count of Participants; unit: Participants] | 11 | 14 | 25
ECOG > 2 [Count of Participants; unit: Participants] — ECOG refers to Eastern Cooperative Oncology Group Performance status. ECOG was recorded as the most recent value documented in the structured ECOG performance status field in the electronic health record at the time of enrollment. The ECOG Performance Status Scale is used to describe patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). ECOG scores are used to help determine a patient's eligibility for clinical trials. ECOG scores range from 0 to 5, with 0 indicating full activity and 5 indicating death.
  Participants | 1 | 0 | 1
Uncontrolled symptoms [Count of Participants; unit: Participants] | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Completion of Palliative Care Visit
Description: Binary outcome (yes/no) measured at the patient level among eligible patients based on the date of documented palliative care encounter
Time Frame: Within 12 weeks of the Index Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 136 | 130
Participants | 11 | 19

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: CRC chart review
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 23/136 | 15/130
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/130
Other Adverse Events (participants affected / at risk) | 0/136 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT05365997/Prot_SAP_000.pdf